CLINICAL TRIAL: NCT02175836
Title: Arrhythmia Prediction Trial and Risk Stratification in Heart Failure Patients - Athens.
Brief Title: Arrhythmia Prediction Trial
Acronym: APRET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, PETROS ARSENOS, MD, PhD, University of Athens
Other Study IDs: 17/25-10-2006; APRET, Athens Medical School (Other: Athens Medical School)
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Myocardial Infarction; Dilated Cardiomyopathy; Heart Failure
Keywords: Arrhythmic Sudden Cardiac Death; Heart Failure; Risk Stratification; Autonomic Nervous System; Heart Rate; Repolarization
MeSH Terms: conditions — Myocardial Infarction; Cardiomyopathy, Dilated; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SCD possitive versus SCD negative group: The total Heart Failure patients subgroup experiencing Sudden Cardiac Death surrogate end-points during follow up versus the patients subgroup that is free from Sudden Cardiac Death surrogate end-points.

SUMMARY:
Patients with Ischaemic and Dilated Cardiomyopathy, face an increased risk for Arrhythmic Sudden Cardiac Death. The purpose of this study is to estimate the performance of Modern Non-Invasive Indices and the performance of Programmed Ventricular Stimulation in Sudden Cardiac Death Prediction.

DETAILED DESCRIPTION:
Sudden Cardiac Death (SCD) threatens survival of Coronary Artery Disease and Dilated Cardiomyopathy patients with Heart Failure. Discovering efficient SCD risk stratification markers is of high importance. In this study, heart failure patients will be risk stratified with indices from the Myocardial substrate (QRS, fragmented QRS, Late potentials, LVEF), indices from the Repolarization status (QT duration, QT rate corrected , QT dispersion, QT/RR, T wave Amplitude Variability, T wave alternans, QT Variability Index), indices from the Autonomic Nervous System function [ Heart Rate variability, Heart rate Turbulence, Deceleration Capacity (DC) , DC sign of fraction, Beat to Beat DC, Non linear indices of Heart Rate Dynamics], the Non sustained ventricular tachycardia and Ventricular extrasystolic activity and the Circadian Properties of Heart Rate observed during Ambulatory Monitoring. Furthermore Programmed Ventricular Stimulation will be used. High resolution 30 min ECG recordings will performed for further indices research and development. All the Arrhythmic Risk Stratifiers will be analysed and their performance for Sudden Cardiac Death Prediction and for Total Mortality will be estimated according the follow up.

ELIGIBILITY:
Inclusion Criteria:

* Myocardial Infarction
* Dilated Cardiomyopathy
* Sinus rhythm

Exclusion Criteria:

* Malignant diseases seriously affecting the survival
* Conditions/diseases affecting the Autonomic Nervous System's function
* Dementia
* Alcoholism
* Psychiatric diseases
* Addiction

Ages: 20 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart Failure Patients with Myoacardial Infarction and Dilated Cardiomyopathy maintaining sinus rhyhtm.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2007-10; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Sudden Cardiac Death surrogates: 1.Clinical Ventricular Tachyarrhythmia, 2.ICD's appropriate activation, 3.Confirmed Sudden Cardiac Death | 2007-2019 (12 years)

SECONDARY OUTCOMES:
Total Mortality | 2007-2019 (12 years)

CONTACTS AND LOCATIONS:
Overall Officials: Petros Arsenos, MD, PhD, Principal Investigator — First Department of Cardiology, Medical School, National & Kapodistrian University of Athens, Greece
Locations (1):
- First Department of Cardiology, Medical School, National & Kapodistrian University of Athens, Athens, Greece

REFERENCES:
- [Background] Mirowski M, Mower MM, Langer A, Heilman MS, Schreibman J. A chronically implanted system for automatic defibrillation in active conscious dogs. Experimental model for treatment of sudden death from ventricular fibrillation. Circulation. 1978 Jul;58(1):90-4. doi: 10.1161/01.cir.58.1.90. PMID 647893
- [Background] Moss AJ, Zareba W, Hall WJ, Klein H, Wilber DJ, Cannom DS, Daubert JP, Higgins SL, Brown MW, Andrews ML; Multicenter Automatic Defibrillator Implantation Trial II Investigators. Prophylactic implantation of a defibrillator in patients with myocardial infarction and reduced ejection fraction. N Engl J Med. 2002 Mar 21;346(12):877-83. doi: 10.1056/NEJMoa013474. Epub 2002 Mar 19. PMID 11907286
- [Background] Bauer A, Barthel P, Schneider R, Ulm K, Muller A, Joeinig A, Stich R, Kiviniemi A, Hnatkova K, Huikuri H, Schomig A, Malik M, Schmidt G. Improved Stratification of Autonomic Regulation for risk prediction in post-infarction patients with preserved left ventricular function (ISAR-Risk). Eur Heart J. 2009 Mar;30(5):576-83. doi: 10.1093/eurheartj/ehn540. Epub 2008 Dec 23. PMID 19109245
- [Background] Arsenos P, Gatzoulis KA, Dilaveris P, Gialernios T, Sideris S, Lazaros G, Archontakis S, Tsiachris D, Kartsagoulis E, Stefanadis C. The rate-corrected QT interval calculated from 24-hour Holter recordings may serve as a significant arrhythmia risk stratifier in heart failure patients. Int J Cardiol. 2011 Mar 3;147(2):321-3. doi: 10.1016/j.ijcard.2010.12.076. Epub 2011 Jan 15. No abstract available. PMID 21239068
- [Background] Gatzoulis KA, Vouliotis AI, Tsiachris D, Salourou M, Archontakis S, Dilaveris P, Gialernios T, Arsenos P, Karystinos G, Sideris S, Kallikazaros I, Stefanadis C. Primary prevention of sudden cardiac death in a nonischemic dilated cardiomyopathy population: reappraisal of the role of programmed ventricular stimulation. Circ Arrhythm Electrophysiol. 2013 Jun;6(3):504-12. doi: 10.1161/CIRCEP.113.000216. Epub 2013 Apr 15. PMID 23588627
- [Background] Arsenos P, Gatzoulis KA, Gialernios T, Dilaveris P, Tsiachris D, Archontakis S, Vouliotis AI, Raftopoulos L, Manis G, Stefanadis C. Elevated nighttime heart rate due to insufficient circadian adaptation detects heart failure patients prone for malignant ventricular arrhythmias. Int J Cardiol. 2014;172(1):e154-6. doi: 10.1016/j.ijcard.2013.12.075. Epub 2013 Dec 28. No abstract available. PMID 24411917
- [Background] Gatzoulis KA, Archontakis S, Dilaveris P, Tsiachris D, Arsenos P, Sideris S, Stefanadis C. Ventricular arrhythmias: from the electrophysiology laboratory to clinical practice. Part I: malignant ventricular arrhythmias. Hellenic J Cardiol. 2011 Nov-Dec;52(6):525-35. No abstract available. PMID 22143016
- [Background] Gatzoulis KA, Tsiachris D, Dilaveris P, Archontakis S, Arsenos P, Vouliotis A, Sideris S, Trantalis G, Kartsagoulis E, Kallikazaros I, Stefanadis C. Implantable cardioverter defibrillator therapy activation for high risk patients with relatively well preserved left ventricular ejection fraction. Does it really work? Int J Cardiol. 2013 Aug 20;167(4):1360-5. doi: 10.1016/j.ijcard.2012.04.005. Epub 2012 Apr 24. PMID 22534047
- [Background] Huikuri HV, Makikallio TH, Raatikainen MJ, Perkiomaki J, Castellanos A, Myerburg RJ. Prediction of sudden cardiac death: appraisal of the studies and methods assessing the risk of sudden arrhythmic death. Circulation. 2003 Jul 8;108(1):110-5. doi: 10.1161/01.CIR.0000077519.18416.43. No abstract available. PMID 12847054
- [Background] Makikallio TH, Barthel P, Schneider R, Bauer A, Tapanainen JM, Tulppo MP, Schmidt G, Huikuri HV. Prediction of sudden cardiac death after acute myocardial infarction: role of Holter monitoring in the modern treatment era. Eur Heart J. 2005 Apr;26(8):762-9. doi: 10.1093/eurheartj/ehi188. Epub 2005 Mar 18. PMID 15778204
- [Background] Wellens HJ, Schwartz PJ, Lindemans FW, Buxton AE, Goldberger JJ, Hohnloser SH, Huikuri HV, Kaab S, La Rovere MT, Malik M, Myerburg RJ, Simoons ML, Swedberg K, Tijssen J, Voors AA, Wilde AA. Risk stratification for sudden cardiac death: current status and challenges for the future. Eur Heart J. 2014 Jul 1;35(25):1642-51. doi: 10.1093/eurheartj/ehu176. Epub 2014 May 5. PMID 24801071
- [Background] Myerburg RJ. Sudden cardiac death: exploring the limits of our knowledge. J Cardiovasc Electrophysiol. 2001 Mar;12(3):369-81. doi: 10.1046/j.1540-8167.2001.00369.x. PMID 11291815
- [Background] Gomes JA, Cain ME, Buxton AE, Josephson ME, Lee KL, Hafley GE. Prediction of long-term outcomes by signal-averaged electrocardiography in patients with unsustained ventricular tachycardia, coronary artery disease, and left ventricular dysfunction. Circulation. 2001 Jul 24;104(4):436-41. doi: 10.1161/hc2901.093197. PMID 11468206
- [Background] Merchant FM, Zheng H, Bigger T, Steinman R, Ikeda T, Pedretti RF, Salerno-Uriarte JA, Klersy C, Chan PS, Bartone C, Hohnloser SH, Ruskin JN, Armoundas AA. A combined anatomic and electrophysiologic substrate based approach for sudden cardiac death risk stratification. Am Heart J. 2013 Oct;166(4):744-52. doi: 10.1016/j.ahj.2013.06.023. Epub 2013 Sep 18. PMID 24093856
- [Background] Schwartz PJ, Wolf S. QT interval prolongation as predictor of sudden death in patients with myocardial infarction. Circulation. 1978 Jun;57(6):1074-7. doi: 10.1161/01.cir.57.6.1074. PMID 639227
- [Background] Exner DV, Kavanagh KM, Slawnych MP, Mitchell LB, Ramadan D, Aggarwal SG, Noullett C, Van Schaik A, Mitchell RT, Shibata MA, Gulamhussein S, McMeekin J, Tymchak W, Schnell G, Gillis AM, Sheldon RS, Fick GH, Duff HJ; REFINE Investigators. Noninvasive risk assessment early after a myocardial infarction the REFINE study. J Am Coll Cardiol. 2007 Dec 11;50(24):2275-84. doi: 10.1016/j.jacc.2007.08.042. Epub 2007 Nov 26. PMID 18068035
- [Background] Schwartz PJ. The autonomic nervous system and sudden death. Eur Heart J. 1998 Jun;19 Suppl F:F72-80. PMID 9651739
- [Background] Bauer A, Barthel P, Muller A, Ulm K, Huikuri H, Malik M, Schmidt G. Risk prediction by heart rate turbulence and deceleration capacity in postinfarction patients with preserved left ventricular function retrospective analysis of 4 independent trials. J Electrocardiol. 2009 Nov-Dec;42(6):597-601. doi: 10.1016/j.jelectrocard.2009.07.013. PMID 19853731
- [Background] De Ferrari GM, Rordorf R, Frattini F, Petracci B, De Filippo P, Landolina M. Predictive value of programmed ventricular stimulation in patients with ischaemic cardiomyopathy: implications for the selection of candidates for an implantable defibrillator. Europace. 2007 Dec;9(12):1151-7. doi: 10.1093/europace/eum230. Epub 2007 Oct 17. PMID 17947251
- [Background] Huikuri HV, Raatikainen MJ, Moerch-Joergensen R, Hartikainen J, Virtanen V, Boland J, Anttonen O, Hoest N, Boersma LV, Platou ES, Messier MD, Bloch-Thomsen PE; Cardiac Arrhythmias and Risk Stratification after Acute Myocardial Infarction study group. Prediction of fatal or near-fatal cardiac arrhythmia events in patients with depressed left ventricular function after an acute myocardial infarction. Eur Heart J. 2009 Mar;30(6):689-98. doi: 10.1093/eurheartj/ehn537. Epub 2009 Jan 20. PMID 19155249
- [Background] Gatzoulis KA, Archontakis S, Dilaveris P, Tsiachris D, Arsenos P, Sideris S, Stefanadis C. Ventricular arrhythmias: from the electrophysiology laboratory to clinical practice. Part II: potentially malignant and benign ventricular arrhythmias. Hellenic J Cardiol. 2012 May-Jun;53(3):217-33. No abstract available. PMID 22653247
- [Background] Arsenos P, Gatzoulis K, Manis G, Gialernios T, Dilaveris P, Tsiachris D, Archontakis S, Kartsagoulis E, Mytas D, Stefanadis C. Decreased scale-specific heart rate variability after multiresolution wavelet analysis predicts sudden cardiac death in heart failure patients. Int J Cardiol. 2012 Feb 9;154(3):358-60. doi: 10.1016/j.ijcard.2011.11.007. Epub 2011 Nov 30. No abstract available. PMID 22133464
- [Background] Arsenos P, Gatzoulis K, Dilaveris P, Manis G, Tsiachris D, Archontakis S, Vouliotis AI, Sideris S, Stefanadis C. Arrhythmic sudden cardiac death: substrate, mechanisms and current risk stratification strategies for the post-myocardial infarction patient. Hellenic J Cardiol. 2013 Jul-Aug;54(4):301-15. No abstract available. PMID 23912922
- See also: Related Info — http://www.researchgate.net/profile/Petros_Arsenos?ev=hdr_xprf